CLINICAL TRIAL: NCT01829399
Title: Control of Tourniquet Pain With an Axillary Ring of Subcutaneous Local Anesthetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-2373
Record Dates: First submitted 2013-03-25; First posted 2013-04-11 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Application Site Discomfort; Medical Device Discomfort
Keywords: Tourniquet pain; Subcutaneous axillary local anesthetic; ability to tolerate tourniquet discomfort.
MeSH Terms: interventions — Bupivacaine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injected with Bupivacaine (Experimental): A subcutaneous axillary ring of 10 to 15 mL of 0.25% Bupivacaine with epinephrine 1:200,000 will be injected in the arm 15 minutes prior to tourniquet inflation.
  Interventions: Drug: Bupivacaine with Epinephrine
- Injected with saline (Sham Comparator): A subcutaneous axillary ring of 10 to 15 mL of normal saline will be injected in the arm 15 minutes prior to tourniquet inflation.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine with Epinephrine — 10-15 mL 0.25% Bupivicaine with epinephrine 1:200,000 subcutaneous axillary ring
  Other Names: Marcaine, Exparel, Sensorcaine
  Arms: Injected with Bupivacaine
Drug: Normal Saline
  Other Names: Placebo
  Arms: Injected with saline

SUMMARY:
Purpose: Even with excellent regional anesthesia of the upper extremity, tourniquet (Tq) pain from an upper arm Tq can limit the ability to use regional anesthesia as the primary anesthetic for surgical procedures on the upper extremity. The aim of this study is to determine whether a subcutaneous ring of local anesthetic on the inner aspect of the upper arm just distal to axillary crease will significantly diminish Tq pain. If it does, peripheral nerve blocks distal to the Tq (i.e., nerve blocks at the elbow) could be used as the primary anesthetic for surgery of the hand and forearm. These distal peripheral nerve blocks have fewer complications than brachial plexus blocks performed at higher levels, and, postoperatively, the patient has better control of his or her arm when distal nerve blocks are used.

Procedures (methods): This is a prospective, cross-over study to examine the effectiveness of an upper arm Subcutaneous ring of local anesthetic alone in relieving Tq pain. This Subcutaneous ring of local anesthetic is often referred to as "Intercostobrachial nerve block" or "Subcutaneous ring anesthesia (SRA)." Twenty volunteers will be randomized into four groups of 5 participants each. During the initial experiment, the first group will be given SRA with 10-15 mL of 0.25% Bupivacaine with Epinephrine 1:200,000 on their dominant arm, the second group will be given SRA with 10-15 mL of 0.25% Bupivacaine with Epinephrine 1:200,000 on their non-dominant arm, the third group will be given "sham" SRA with saline on their dominant arm, and the fourth group will be given "sham" SRA with saline on their non-dominant arm. 15 minutes after SRA, a Tq will be applied to the arm with the subcutaneous injection and it will be inflated to 100 mm Hg above the subject's baseline systolic blood pressure. We will monitor heart rate, blood pressure (opposite arm) and pain (0 to 10 VAS) every 5 minutes. Each Tq will be released when the subject requests deflation or when 1 hour of Tq time has elapsed, whichever occurs first. The subject's discomfort level (VAS) just prior to deflation will be recorded. Since Tq pressure alone can inhibit nerve function, we will monitor motor and sensory function distal to the Tq every 10 minutes during Tq inflation and for 30 minutes after Tq deflation. One to two weeks after this initial study, the same 20 subjects will receive SRA on the same arm and the same parameters will be measured. The 10 subjects who received 0.25% Bupivacaine the first time will receive Normal Saline, and the 10 subjects who received Normal Saline the first time will receive 0.25% Bupivacaine. In this way, each subject will act as his or her own control.

ELIGIBILITY:
Inclusion Criteria: Volunteers will be eligible for the study if they meet all of the below criteria;

* American Society of Anesthesiologists (ASA) classification I or II
* 18 years of age to a maximum of 70 years of age

Exclusion criteria:

* Pre-existing parasthesia or neuropathy of any kind
* History of excessive alcohol consumption (> three drinks per night)
* Take analgesics on a regular basis
* History of any drug abuse
* Baseline systolic blood pressure ≥ 150
* Baseline diastolic blood pressure ≥ 85
* BMI ≥ 30 Pregnancy Allergic reaction to local anesthetic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall F Coombs, M.D., Principal Investigator — University of NC at Chapel Hill Dept. of Anesthesiology
Locations (1):
- University of North Carolina at Chapel Hill Medical Center, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine Ring 1st Visit, Saline Ring 2nd Visit: Participants received a subcutaneous axillary ring injection with 0.25% Bupivacaine with epinephrine 1:200.000 on the first visit and a subcutaneous axillary ring injection with saline on the second visit.
- Saline Ring 1st Visit, Bupivacaine Ring 2nd Visit: Participants received a subcutaneous axillary ring injection with normal saline on the first visit and a subcutaneous axillary ring injection with 0.25% Bupivacaine with epinephrine 1:200.000 on the second visit.
Period: Visit 1
Arm/Group | Bupivacaine Ring 1st Visit, Saline Ring 2nd Visit | Saline Ring 1st Visit, Bupivacaine Ring 2nd Visit
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Visit 2 (One Month Later)
Arm/Group | Bupivacaine Ring 1st Visit, Saline Ring 2nd Visit | Saline Ring 1st Visit, Bupivacaine Ring 2nd Visit
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bupivacaine Ring 1st Visit, Saline Ring 2nd Visit: On the first visit, subcutaneous axillary ring of 10 to 15 ml of 0.25% Bupivacaine with epinephrine 1:200,000 was injected 15 minutes prior to tourniquet inflation. On the second visit, a subcutaneous axillary ring of 10 to 15 ml of saline was injected 15 minutes prior to tourniquet inflation.
- Saline Ring 1st Visit, Bupivacaine Ring 2nd Visit: On the first visit, a subcutaneous axillary ring of 10 to 15 mL of normal saline was injected 15 minutes prior to tourniquet inflation. On the second visit, a subcutaneous axillary ring of 10 to 15 ml of 0.25% Bupivacaine with epinephrine 1:200,000 was injected 15 minutes prior to tourniquet inflation.
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Ring 1st Visit, Saline Ring 2nd Visit | Saline Ring 1st Visit, Bupivacaine Ring 2nd Visit | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (10.0) | 32.3 (10.5) | 32.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Arm Dominance [Number; unit: participants] — Since clinical tourniquet application may be on the patients dominant arm or non-dominant arm, participants were stratified according to dominant or non-dominant arm in order to make the results of this study more generalisable.
  participants
    Dominant Arm | 6 | 6 | 12
    Non-Dominant Arm | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Time in Minutes That Tq Remained Inflated
Description: 15 minutes after either Bupivacaine or placebo injection, Tq was inflated to 100 mm Hg over subjects systolic blood pressure. When the subject found the Tq too uncomfortable, the Tq was deflated and the time documented. Approximately one month later, each subject had the opposite injection of either placebo or Bupivacaine on the same arm, and the duration of Tq inflation was again measured. Due to a strong crossover effect, only the data assessed from the first intervention was analyzed.
Time Frame: Tq was inflated 15 minutes after injection of Bupivacaine or placebo and remained inflated until subject could no longer tolerate it. Maximum allowable inflation time per session was 60 minutes.
Measure: Mean (95% Confidence Interval); unit: Minutes
Groups:
- Bupivacaine Axillary Ring on 1st Visit: Participants received a subcutaneous axillary ring injection with 0.25% Bupivacaine with epinephrine 1:200.000.
- Saline Axillary Ring on 1st Visit (Control Group): Participants received a subcutaneous axillary ring injection with normal saline.
Arm/Group | Bupivacaine Axillary Ring on 1st Visit | Saline Axillary Ring on 1st Visit (Control Group)
Number analyzed (Participants) | 12 | 12
Minutes | 30.5 [26.1 to 35.0] | 22.4 [18.0 to 26.9]

2. Secondary Outcome: Pain Score at Time of Tq Deflation
Description: A visual analog pain score (VAS) from 0 to 10 was assessed at the time of Tq deflation. 0 indicating no pain, and 10 indicating the worst possible pain. All participants requested deflation prior to the maximum allowable 60 minutes, Subjects were instructed to request deflation at the same degree of discomfort for each visit. Due to a strong crossover effect, only the data assessed from the first intervention was analyzed.
Time Frame: Tq will be deflated upon subject's request. VAS is assessed at time of deflation for degree of discomfort prompting deflation request, up to 60 minutes post intervention.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Bupivacaine Ring 1st Visit: On the first visit, a subcutaneous axillary ring of 10 to 15 mL of 0.25% Bupivacaine with epinephrine 1:200,000 was injected 15 minutes prior to tourniquet inflation.
- Saline Axillary Ring on 1st Visit (Control Group): On the first visit, a subcutaneous axillary ring of 10 to 15 mL of normal saline was injected 15 minutes prior to tourniquet inflation.
Arm/Group | Bupivacaine Ring 1st Visit | Saline Axillary Ring on 1st Visit (Control Group)
Number analyzed (Participants) | 12 | 12
scores on a scale | 6.1 [5.2 to 7.1] | 5.0 [4.0 to 5.9]

ADVERSE EVENTS:
Groups:
- Bupivacaine Axillary Ring: Participants received a subcutaneous axillary ring injection with 0.25% Bupivacaine with epinephrine 1:200.000
- Saline Axillary Ring (Control Group): Participants received a subcutaneous axillary ring injection with normal saline
Arm/Group | Bupivacaine Axillary Ring | Saline Axillary Ring (Control Group)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Originally this was designed as a crossover study. However, there was a very strong crossover effect which invalidated the results from the second series of injections. Therefore, we have only analyzed the data from the first visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes